CLINICAL TRIAL: NCT04446130
Title: A Phase 3, Open Label, Single Arm, Multi-Center Study to Evaluate the Efficacy and Safety of Decitabine Combined With HAAG Regimen in Newly Diagnosed ETP-ALL/LBL, T/M-MPAL and ALL/LBL With Myeloid or Stem Cell Markers Patients
Brief Title: Study of Decitabine Combined With HAAG Regimen in Newly Diagnosed ETP-ALL/LBL, T/M-MPAL and ALL/LBL With Myeloid or Stem Cell Markers Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Henan Cancer Hospital (Other Government); Shandong Provincial Hospital (Other Government); Shenzhen People's Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Changzhou No.2 People's Hospital (Other); The Second People's Hospital of Huai'an (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAC-HAAG-03
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Induction Chemotherapy; Acute T-Lymphocytic Leukemia; T-cell Lymphoblastic Lymphoma Leukemia; T-cell/Myeloid Mixed Phenotype Acute Leukemia
Keywords: T-ALL/LBL; T/M-MPAL; Decitabine combined with HAAG
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decitabine combined with HAAG Regimen (Experimental): This cohort will determine the safety and efficacy of decitabine combined with HAAG regimen in the newly diagnosed T-ALL/LBL and T/M-MPAL patients.
  Interventions: Drug: Decitabine combined with HAAG Regimen

INTERVENTIONS:
Drug: Decitabine combined with HAAG Regimen — Decitabine :20mg/m2/d,d1~5, intravenous infusion; Homoharringtonine :1mg/d,d3~16,intravenous infusion; Aclarubicin :10mg/d, d3~d10, intravenous infusion; Cytarabine :10mg/m2,q12h,d3-16, subcutaneous injection; Granulocyte colony-stimulating factor (G-CSF): 50-300μg/d (when WBC counts are less than 20×10^9/L ),subcutaneous injection

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of decitabine combined with HAAG regimen in the treatment of newly diagnosed patients with ETP-ALL/LBL, T/M-MPAL and ALL/LBL with myeloid or stem cell markers.

DETAILED DESCRIPTION:
This is a phase 3, open label, single arm, multi-center study in newly diagnosed ETP-ALL/LBL, T/M-MPAL and ALL/LBL patients who have myeloid or stem cell markers. The patients will receive decitabine combined with HAAG regimen in the induction treatment. The patients who respond to induction chemotherapy will undergo consolidation chemotherapy, and an optional allogeneic hematopoietic stem cell transplantation and post-transplantation maintenance treatment with decitabine according to patient's wishes.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed ETP-ALL/LBL, T/M-MPAL according to the 2016 revision to the WHO classification of myeloid neoplasms and acute leukemia, and T-ALL/LBL with one or more of the myeloid or stem cell markers (CD34, CD117, HLADR, CD13, CD33, CD11b or CD65) on at least 25% of lymphoblasts.
2. Age 15-60.
3. Eastern Cooperative Oncology Group (ECOG) score: 0-2.
4. No history of previous chemotherapy or target therapy.
5. Provide informed consent.

Exclusion Criteria:

1. Patients with another malignant disease.
2. Patients has participated in or participating in other clinical trials.
3. Patients with uncontrolled active infection.
4. Patients with left ventricular ejection fraction < 0.5 by echocardiography or grade III/IV cardiovascular dysfunction according to the New York Heart Association Classification.
5. Patients with aspartate aminotransferase or glutamic-pyruvic transaminase > 3x upper limit of normal or bilirubin > 2.0 mg/dL.
6. Patients with creatinine clearance rate < 50ml/min.
7. Patients with active hepatitis B or hepatitis C infection.
8. Patients with HIV infection.
9. Patients with active tuberculosis infection.
10. Patients with uncontrolled active bleeding.
11. Patients with a history of allergy to experimental drugs.
12. Patients with other commodities that the investigators considered not suitable for the enrollment.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Day 28-35 of induction course
  ORR includes complete remission (CR), CR with incomplete hematologic recovery (CRi) and partial remission (PR). CR was defined as < 5% bone marrow blasts in an aspirate with spicules and independent of transfusions; CRi: was defined as<5% bone marrow blasts, either ANC<1×10^9/L or platelets<100×10^9/L, transfusion independence but with persistence of cytopenia; PR was defined as decrease of at least 50% in the percentage of blasts to 5-25% in the bone marrow aspirate and the normalization of blood counts.

SECONDARY OUTCOMES:
Overall survival (OS) | 4 years
  time from randomization to death from any cause
Leukemia-free survival (LFS) | 4 years
  time from randomization to the first relapse or death
Cumulative incidence of relapse(CIR) | 4 years
  time from achievement of a remmission to the first relapse
Number of adverse events | 3 years
  adverse events are evaluated with CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China